CLINICAL TRIAL: NCT03332667
Title: A Phase I Study of 131I-MIBG With Dinutuximab +/- Vorinostat for Relapsed/Refractory Neuroblastoma
Brief Title: MIBG With Dinutuximab +/- Vorinostat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Collaborators: United Therapeutics (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NANT2017-01; 2P01CA217959 (NIH)
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — 3-Iodobenzylguanidine; dinutuximab; Vorinostat; sargramostim; Potassium Iodide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A DL1 (Experimental): Patients will receive 131I-MIBG on day 1 at 12 mCi/kg/dose. Dinutuximab is given intravenously on days 8-11 and 29-32 of therapy at 17.5 mg/m2/dose. Patient will receive GM-CSF on days 8-17 and 29-38 at 250 mcg/m2. All patients will receive autologous hematopoietic stem cell infusion on day 15 (+/- 2) of therapy
  Interventions: Radiation: 131I-MIBG; Drug: Dinutuximab; Drug: Sargramostim; Drug: Potassium Iodide
- Cohort A DL2 (Experimental): Patients will receive 131I-MIBG on day 1 at 15 mCi/kg/dose. Dinutuximab is given intravenously on days 8-11 and 29-32 of therapy at 17.5 mg/m2/dose. Patient will receive GM-CSF on days 8-17 and 29-38 at 250 mcg/m2. All patients will receive autologous hematopoietic stem cell infusion on day 15 (+/- 2) of therapy
  Interventions: Radiation: 131I-MIBG; Drug: Dinutuximab; Drug: Sargramostim; Drug: Potassium Iodide
- Cohort A DL3 (Experimental): Patients will receive 131I-MIBG on day 1 at 18 mCi/kg/dose. Dinutuximab is given intravenously on days 8-11 and 29-32 of therapy at 17.5 mg/m2/dose. Patient will receive GM-CSF on days 8-17 and 29-38 at 250 mcg/m2. All patients will receive autologous hematopoietic stem cell infusion on day 15 (+/- 2) of therapy
  Interventions: Radiation: 131I-MIBG; Drug: Dinutuximab; Drug: Sargramostim; Drug: Potassium Iodide
- Cohort B DL4 (Experimental): Vorinostat will be given on days 0-13 at 180 mg/m2/dose. Patients will receive 131I-MIBG on day 1 at 18 mCi/kg/dose. Dinutuximab is given intravenously on days 8-11 and 29-32 of therapy at 17.5 mg/m2/dose. Patient will receive GM-CSF on days 8-17 and 29-38 at 250 mcg/m2. All patients will receive autologous hematopoietic stem cell infusion on day 15 (+/- 2) of therapy
  Interventions: Radiation: 131I-MIBG; Drug: Dinutuximab; Drug: Vorinostat; Drug: Sargramostim; Drug: Potassium Iodide

INTERVENTIONS:
Radiation: 131I-MIBG — Patients will receive 131I-MIBG on day 1. 131I-MIBG dose will be based on the dose level assigned at the time of patient registration
  Other Names: 131I-Metaiodobenzylguanidine; Iobenguane sulfate; m-Iodobenzylguanidine sulfate; MIBG
Drug: Dinutuximab — Dinutuximab is given intravenously on days 8-11 and 29-32 of therapy. Dinutuximab dose will be based on the dose level assigned at the time of patient registration.
  Other Names: Chimeric Monoclonal Antibody 14.18; MAB Ch 14.18; Unituxin; Ch14.18
Drug: Vorinostat — Vorinostat will be given on day 0-13. Vorinostat dose will be based on the dose level assigned at the time of patient registration.
  Other Names: Zolina
  Arms: Cohort B DL4
Drug: Sargramostim — Sargramostim (GM-CSF) will be given on day 8-17 at 250 mcg/m^2
Drug: Potassium Iodide — Potassium iodide will be given by mouth at a dose of 6mg/kg 8-12 hours prior to infusion of 131I-MIBG on Day 1 and then 1mg/kg/dose by mouth starting 4-6 hours after completion of MIBG infusion and continuing every 4 hours on protocol days 1-7 and then 1mg/kg/dose by mouth once daily on protocol days 8-45

SUMMARY:
131I-Metaiodobenzylguanidine (131I-MIBG) is one of the most effective therapies utilized for neuroblastoma patients with refractory or relapsed disease. In this pediatric phase 1 trial, 131I-MIBG will be given in combination with dinutuximab, a chimeric 14.18 monoclonal antibody. This study will utilize a traditional Phase I rolling 6 dose escalation design to determine a recommended phase 2 pediatric dose. An expansion cohort of an additional 6 patients will then be enrolled. If tolerable, vorinostat will then be added to the third dose level. A 6 patient expansion cohort may then be enrolled.

DETAILED DESCRIPTION:
131I-Metaiodobenzylguanidine (131I-MIBG) is one of the most effective therapies utilized for neuroblastoma patients with refractory or relapsed disease. Data from pre-clinical and adult studies suggest that radiation can enhance the efficacy of immunotherapy and targeted therapies such as dinutuximab. This first pediatric phase 1 trial of 131I-MIBG in combination with dinutuximab and vorinostat aims to determine the recommended phase 2 pediatric dose of these three therapies in combination.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have evidence of MIBG uptake into tumor at ≥ 1 site (bone or soft tissue) within 28 days prior to study entry and subsequent to any intervening therapy.
2. Patients must have a diagnosis of neuroblastoma either by histologic verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines.
3. Patients must have a history of high-risk neuroblastoma according to COG risk classification at the time of study registration. Patients who were initially considered low or intermediate-risk, but then reclassified as high-risk are also eligible.
4. All patients must have at least one of the following

   1. Recurrent/progressive disease: after the diagnosis of high risk neuroblastoma at any time prior to enrollment regardless of response to frontline therapy
   2. No prior history of recurrent/progressive disease since the diagnosis of high risk neuroblastoma b1) Refractory disease- a best overall response of no response/stable disease since diagnosis of high risk neuroblastoma and at least 4 cycles of induction therapy. No prior history of recurrent/progressive disease since the diagnosis of high risk neuroblastoma.

      b2) Persistent disease- a best overall response of no partial response since diagnosis of high risk neuroblastoma and at least 4 cycles of induction therapy. No prior history of recurrent/progressive disease since the diagnosis of high risk neuroblastoma.
5. Patients must have at least ONE of the following (lesions may have received prior radiation therapy as long as they meet the other criteria listed below):

   a) For recurrent/progressive or refractory disease, at least one MIBG avid bone site.

   b) For persistent disease, if a patient has 3 or more MIBG avid lesions, then no biopsy is required. If a patients has only 1 or 2 MIBG avid bone lesion sites then biopsy confirmation of neuroblastoma or ganglioneuroblastoma in at least one MIBG avid site present at the time of enrollment is required to be obtained at any time point prior to enrollment.

   c) For MIBG non-avid tumors, patients must have at least one FDG avid site and a biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma at any time prior to enrollment from at least one FDG-avid site.
6. Any amount of neuroblastoma tumor cells in the bone marrow done at the time of study enrollment based on routine morphology with or without immunocytochemistry in at least one sample from bilateral aspirates and biopsies.
7. At least one soft tissue lesion that meets criteria for a TARGET lesion as defined by:

   a) SIZE: Lesion can be accurately measured in at least one dimension with a longest diameter ≥ 10 mm, or for lymph nodes ≥ 15 mm on short axis. Lesions meeting size criteria will be considered measurable.

   b) In addition to size, a lesion needs to meet one of the following criteria except for patients with parenchymal CNS lesions which only need to meet size criteria: b1) MIBG avid. For patients with recurrent/progressive or refractory disease, no biopsy is required. For patients with persistent disease only: If a patient has only 1 or 2 MIBG avid lesions sites, then biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one MIBG avid site present at time of enrollment is required to be obtained. If a patient has 3 or more MIBG avid lesions, then no biopsy is required.

   b2) MIBG non avid tumors: Patients must have at least one FDG avid site and biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one FDG-PET avid site present at the time of enrollment.
8. At least one non-target soft tissue lesion that is not measurable, but had a biopsy positive for neuroblastoma and/or ganglioneuroblastoma or is MIBG avid at any time prior to enrollment.
9. Patients must have a life expectancy of at least 12 weeks and a Lansky (≤16 years) or Karnofsky (>16 years) score of at least 50.
10. Prior Therapy 1. Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to study registration.

2. Patients must not have received the therapies indicated below after disease evaluation or within the specified time period prior to registration on this study as follows:

1. Myelosuppressive chemotherapy: must not have received within 2 weeks prior to registration.

2. Biologic anti-neoplastics- agents not known to be associated with reduced platelet or ANC counts (including retinoids): must not have received within 7 days prior to registration.

3. Monoclonal antibodies: must have received last dose at least 7 days or 3 half-lives whichever is longer, but no longer than 30 days (with recovery of any associated toxicities), prior to protocol therapy.

4. Cellular Therapy (e.g. modified T cells, NK cells, dentritic cells etc.): must not have received within 3 weeks and resolution of all toxicities.

5. Radiation: must not have received small port radiation within 7 days prior to registration.

6. Hematopoietic Stem Cell Transplant: 7. IVIG 8. Therapeutic MIBG 9. Investigational medicines covered under another IND 10. Medications interfering with MIBG uptake 11. Medications that prolong QTc (Part B only) 12. Valproic acid (Part B only) 11) All patients must have adequate organ function defined as:

- Hematological Function:

1. Absolute Phagocyte count (APC= neutrophils and monocytes): ≥ 1000/µL
2. Absolute Neutrophil count: ≥750/µL
3. Absolute Lymphocyte count ≥ 500/µL
4. Platelet count: ≥ 50,000/µL, transfusion independent (no platelet transfusions within 1 week)
5. Hemoglobin ≥ 10 g/dL (may transfuse)
6. Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria above.

   * Renal Function: Age-adjusted serum creatinine ≤ to 1.5 x normal for age/gender OR creatinine clearance or GFR greater than or equal to 60 cc/min/1.73m2
   * Liver Function: Total bilirubin ≤ 1.5 x normal for age, AND SGPT (ALT) 135 and SGOT (AST) ≤ 3 x upper limit of normal. Sinusoidal obstruction syndrome (SOS) if present, must be stable or improving clinically
   * Cardiac Function: Normal ejection fraction documented by either echocardiogram or radionuclide MUGA evaluation OR Normal fractional shortening documented by echocardiogram
   * Pulmonary Function: No dyspnea at rest, no oxygen requirement.

     12) Reproductive Status: All post-menarchal females must have a negative beta-HCG. Males and females of reproductive age and childbearing potential must use effective contraception for the duration of their participation.

     13) Patients with other ongoing serious medical issues must be approved by the study chair prior to registration.

     14) Autologous peripheral blood stem cells (PBSC)•The minimum dose for peripheral blood stem cells is 2.0 x 106viable CD34+ cells/kg. Patients who do not meet this minimum requirement for available PBSCs are not eligible. •Only un-purged stem cells are allowed unless a center has separate FDA approval for infusion of purged stem cells. •For patients whose body weight exceeds ideal body weight (IBW) by more than 20%, adjusted body weight may be used for the calculation of PBSC dose 15) Physician deems that there is reasonable ability to obtain vorinostat via commercial supply (Part B Only)

Exclusion Criteria:

* Pregnancy, breast feeding, or unwillingness to use effective contraception during the study.
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
* Patients with disease of any major organ system that would compromise their ability to withstand therapy.
* Patients who have received prior allogeneic stem cell transplant
* Patients who have received prior solid organ transplantation
* Patients must not have received prior total body irradiation
* Prior HDAC inhibitor given in combination with therapeutic 131I-MIBG(Part B only)
* The maximum total allowable dose of 131I-MIBG that can be given per institutional guidelines must be at least 90% of the calculated 131I-MIBG dose or the patient is not eligible.
* Patients who are on hemodialysis.
* Patients with an active or uncontrolled infection.
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C.
* Patient declines participation in NANT 2004-05, the NANT Biology Study
* Patients and/or families who are physically and psychologically unable to cooperate with the radiation safety isolation.
* Patients with a history of having to discontinue anti-GD2 antibody therapy due to toxicity are not eligible.
* Prior anti-GD2 therapy is not otherwise an exclusionary criteria unless it was given in combination with therapeutic 131I-MIBG.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cash, MD, Study Chair — Children's Healthcare of Atlanta; Araz Marachelian, MD, MS, Study Director — Children's Hospital Los Angeles
Locations (12):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children Hospital of Colorado, Aurora, Colorado
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - University of Chicago, Comer Children's Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - C.S Mott Children's Hospital, Ann Arbor, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Healthcare System, Fort Worth, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cash T, Marachelian A, DuBois SG, Chi YY, Baregamyan A, Groshen SG, Jonus HC, Shamirian A, Crowley M, Goodarzian F, Acharya PT, Pawel B, Erbe AK, Shahi A, Zaborek J, Kennedy E, Asgharzadeh S, Villablanca JG, Pinto N, Weiss BD, Mosse YP, Desai AV, Macy ME, Granger M, Vo KT, Sondel PM, Matthay KK, Park JR, Goldsmith KC. Phase I Study of 131I-Metaiodobenzylguanidine With Dinutuximab +/- Vorinostat for Patients With Relapsed or Refractory Neuroblastoma: A New Approaches to Neuroblastoma Therapy Trial. J Clin Oncol. 2025 Aug;43(22):2490-2501. doi: 10.1200/JCO-24-02612. Epub 2025 Jun 23. PMID 40549985

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A DL1: Patients will receive 131I-MIBG on day 1 at 12mCI/kg/dose. Dinutuximab is given intravenously on days 8-11 and 29-32 of therapy at 17mg/m2/dose. Patient will receive GM-CSF on days 8-17 and 29-38 at 250 mcg/m2. All patients will receive autologous hematopoietic stem cell infusion on day 15 (+/- 2) of therapy.
- Cohort A DL2: Patients will receive 131I-MIBG on day 1 at 15mCI/kg/dose. Dinutuximab is given intravenously on days 8-11 and 29-32 of therapy at 17mg/m2/dose. Patient will receive GM-CSF on days 8-17 and 29-38 at 250 mcg/m2. All patients will receive autologous hematopoietic stem cell infusion on day 15 (+/- 2) of therapy.
- Cohort A DL3: 1 at 18mCI/kg/dose. Dinutuximab is given intravenously on days 8-11 and 29-32 of therapy at 17mg/m2/dose. Patient will receive GM-CSF on days 8-17 and 29-38 at 250 mcg/m2. All patients will receive autologous hematopoietic stem cell infusion on day 15 (+/- 2) of therapy.
- Cohort B DL4: Vorinostat will be given on days 0-13 at 180mg/m2/dose. Patients will receive 131I-MIBG on day 1 at 18mCI/kg/dose. Dinutuximab is given intravenously on days 8-11 and 29-32 of therapy at 17mg/m2/dose. Patient will receive GM-CSF on days 8-17 and 29-38 at 250 mcg/m2. All patients will receive autologous hematopoietic stem cell infusion on day 15 (+/- 2) of therapy.
Period: Overall Study
Arm/Group | Cohort A DL1 | Cohort A DL2 | Cohort A DL3 | Cohort B DL4
Started | 6 | 5 | 20 | 14
Completed | 1 | 2 | 6 | 11
Not Completed | 5 | 3 | 14 | 3
Not completed — Adverse Event | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 5 | 1
Not completed — Disease Progression or Relapse | 2 | 1 | 3 | 0
Not completed — Initiation onto Another Anti-Cancer Therapy | 1 | 1 | 3 | 1
Not completed — No Treatment Received | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort A DL3: Patients will receive 131I-MIBG on day 1 at 18mCI/kg/dose. Dinutuximab is given intravenously on days 8-11 and 29-32 of therapy at 17mg/m2/dose. Patient will receive GM-CSF on days 8-17 and 29-38 at 250 mcg/m2. All patients will receive autologous hematopoietic stem cell infusion on day 15 (+/- 2) of therapy.
- Total: Total of all reporting groups
Arm/Group | Cohort A DL1 | Cohort A DL2 | Cohort A DL3 | Cohort B DL4 | Total
Number analyzed (Participants) | 6 | 5 | 20 | 14 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 5 | 19 | 11 | 40
  Between 18 and 65 years | 1 | 0 | 1 | 3 | 5
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 7 | 7 | 18
  Male | 4 | 3 | 13 | 7 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 3 | 1 | 8
  Not Hispanic or Latino | 4 | 2 | 14 | 13 | 33
  Unknown or Not Reported | 1 | 0 | 3 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 2 | 5
  White | 5 | 3 | 12 | 9 | 29
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 2 | 4 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: MTD/RP2D Determination Cohort A
Description: Proportion of patients with Course 1 DLT in Cohort A
Time Frame: All toxicities from enrollment until completion of course 1 (Day 56)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A DL1 | Cohort A DL2 | Cohort A DL3
Number analyzed (Participants) | 4 | 4 | 11
Participants | 0 | 0 | 0

2. Primary Outcome: MTD/RP2D Determination Cohort B
Description: Proportion of patients with Course 1 DLT in Cohort B
Time Frame: All toxicities from enrollment until completion of course 1 (Day 56)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B DL4
Number analyzed (Participants) | 12
Participants | 1

3. Primary Outcome: Describe Non-Hematological Toxicities Cohort A
Description: Proportion of patients with any grade 3 or greater non-hematological toxicities in Cohort A
Time Frame: All toxicities from enrollment through 30 days following end of protocol therapy, up to 5 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A DL2: Patients will receive 131I-MIBG on day 1 at 12mCI/kg/dose. Dinutuximab is given intravenously on days 8-11 and 29-32 of therapy at 17mg/m2/dose. Patient will receive GM-CSF on days 8-17 and 29-38 at 250 mcg/m2. All patients will receive autologous hematopoietic stem cell infusion on day 15 (+/- 2) of therapy.
Arm/Group | Cohort A DL1 | Cohort A DL2 | Cohort A DL3
Number analyzed (Participants) | 6 | 5 | 19
Participants | 5 | 3 | 10

4. Primary Outcome: Describe Non Hematological Toxicities Cohort B
Description: Proportion of patients with any grade 3 or greater non-hematological toxicities in Cohort B
Time Frame: All toxicities from enrollment through 30 days following end of protocol therapy, up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B DL4
Number analyzed (Participants) | 14
Participants | 12

5. Secondary Outcome: Overall Response Cohort A
Description: Proportion of patients evaluable for response with a best overall response of CR/CR-MD/PR for patients in Cohort A
Time Frame: From Day 1 of protocol therapy through 30 days following end of protocol therapy, up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A DL1 | Cohort A DL2 | Cohort A DL3
Number analyzed (Participants) | 6 | 5 | 15
Participants | 2 | 4 | 5

6. Secondary Outcome: Overall Response Cohort B
Description: Proportion of patients evaluable for response with a best overall response of CR/CR-MD/PR for patients in Cohort B
Time Frame: From Day 1 of protocol therapy through 30 days following end of protocol therapy, up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B DL4
Number analyzed (Participants) | 12
Participants | 5

ADVERSE EVENTS:
Time Frame: All adverse events from enrollment through 30 days following end of protocol therapy, up to 5 months
Description: Adverse events were collected through regular investigator assessment and regular laboratory testing.
Arm/Group | Cohort A DL1 | Cohort A DL2 | Cohort A DL3 | Cohort B DL4
All-Cause Mortality (participants affected / at risk) | 4/6 | 1/5 | 12/20 | 5/14
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/5 | 6/20 | 8/14
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 19/20 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A DL1 (N=6) | Cohort A DL2 (N=5) | Cohort A DL3 (N=20) | Cohort B DL4 (N=14)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Jejunal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fever (General disorders) | 0 | 1 | 0 | 2
Pain (General disorders) | 0 | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A DL1 (N=6) | Cohort A DL2 (N=5) | Cohort A DL3 (N=20) | Cohort B DL4 (N=14)
Anemia (Blood and lymphatic system disorders) | 6 | 4 | 16 | 12
BLEEDING (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Methemoglobinemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
GALLOP RHYTHM (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 4
Sinus tachycardia (Cardiac disorders) | 5 | 2 | 9 | 7
Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 2 | 3
EYE DISCHARGE (Eye disorders) | 0 | 0 | 0 | 1
EYE ITCHINESS (Eye disorders) | 0 | 0 | 1 | 0
Periorbital edema (Eye disorders) | 0 | 1 | 1 | 0
REDNESS (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 3 | 6
Constipation (Gastrointestinal disorders) | 4 | 2 | 6 | 6
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 4 | 9
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 2 | 14 | 12
ORAL THRUSH (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 5 | 10 | 12
Disease Progression (General disorders) | 1 | 0 | 0 | 0
Edema face (General disorders) | 0 | 0 | 2 | 1
Edema limbs (General disorders) | 0 | 0 | 1 | 1
Facial pain (General disorders) | 0 | 0 | 2 | 5
Fatigue (General disorders) | 3 | 2 | 5 | 6
Fever (General disorders) | 3 | 3 | 8 | 11
Flu like symptoms (General disorders) | 0 | 0 | 1 | 0
Generalized edema (General disorders) | 0 | 0 | 1 | 1
Injection site reaction (General disorders) | 0 | 1 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1
Pain (General disorders) | 4 | 3 | 10 | 7
Allergic reaction (Immune system disorders) | 0 | 0 | 3 | 0
Anaphylaxis (Immune system disorders) | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1
Conjunctivities (Infections and infestations) | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 2 | 3
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis infective (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Thrush (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 2 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2 | 10 | 11
Alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 11 | 11
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 2 | 6
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 2
Creatinine increased (Investigations) | 0 | 0 | 3 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 2
GGT increased (Investigations) | 0 | 2 | 0 | 0
Hemoglobin increased (Investigations) | 1 | 1 | 1 | 0
INR increased (Investigations) | 2 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 6 | 5 | 16 | 14
Neutrophil count decreased (Investigations) | 5 | 3 | 15 | 13
Platelet count decreased (Investigations) | 5 | 5 | 16 | 13
Thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 0
Weight gain (Investigations) | 0 | 0 | 0 | 1
Weight loss (Investigations) | 1 | 1 | 4 | 5
White blood cell decreased (Investigations) | 6 | 5 | 18 | 13
Anorexia (Metabolism and nutrition disorders) | 2 | 2 | 10 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 2 | 6 | 9
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 4
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 5 | 13 | 12
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 4 | 10 | 12
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 5 | 4 | 6 | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 3 | 4 | 6
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 8 | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 3 | 10 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
JAW PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 4
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 4
Hypersomnia (Nervous system disorders) | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 2
Movements involuntary (Nervous system disorders) | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1
Spasticity (Nervous system disorders) | 0 | 1 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 5 | 3
Anxiety (Psychiatric disorders) | 0 | 1 | 2 | 3
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 1 | 2
Dysuria (Renal and urinary disorders) | 1 | 1 | 1 | 0
FOLEY PAIN (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 2 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 2 | 0 | 2 | 4
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 6 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
RHINOVIRUS OR ENTEROVIRUS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3
DIAPER RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
IRRITATION AT PORT SITE (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
PERINEUM REDNESS & ITCHSING (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 6 | 6
REDNESS FROM RUBBING (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
UNSPECIFIED NON-PRURITIC RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Capillary leak syndrome (Vascular disorders) | 0 | 1 | 1 | 3
Hypertension (Vascular disorders) | 5 | 0 | 5 | 4
Hypotension (Vascular disorders) | 2 | 2 | 7 | 7
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT03332667/Prot_SAP_ICF_000.pdf